CLINICAL TRIAL: NCT01331668
Title: Biobank Renal Transplantation University Hospitals Leuven
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Maarten Naesens, Prof. Dr. Maarten Naesens, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: TRA-UZL-BIOBANK-001
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Kidney Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy material (tissue, RNA, DNA) Peripheral blood samples (serum, plasma, RNA, DNA) Urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- renal allograft donors and recipients: All de novo renal allograft recipients transplanted at the University Hospitals Leuven

SUMMARY:
This study aims to maintain a prospective biobank of human samples obtained from donors and recipients of renal allografts, including biopsy tissue, peripheral blood samples and urine samples.

DETAILED DESCRIPTION:
Clinical data and bio-specimens are prospectively collected and stored for undefined future translational research projects.

ELIGIBILITY:
Inclusion Criteria:

* renal transplant recipients/donors

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All donors and recipients of a kidney transplant at the University Hospitals Leuven
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2004-03; Primary Completion 2099-12 (Estimated); Study Completion 2099-12 (Estimated)

PRIMARY OUTCOMES:
Renal allograft survival | 50 years after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Naesens, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Department of Nephrology and Renal Transplantation - University Hospitals Leuven, Leuven, BE, Belgium

REFERENCES:
- [Background] Naesens M, Heylen L. Intrarenal resistive index after renal transplantation. N Engl J Med. 2014 Feb 13;370(7):677-8. doi: 10.1056/NEJMc1315502. No abstract available. PMID 24521121
- [Result] Kuypers DR, de Jonge H, Naesens M, Vanrenterghem Y. A prospective, open-label, observational clinical cohort study of the association between delayed renal allograft function, tacrolimus exposure, and CYP3A5 genotype in adult recipients. Clin Ther. 2010 Nov;32(12):2012-23. doi: 10.1016/j.clinthera.2010.11.010. PMID 21118736
- [Result] Kuypers DR, Naesens M, de Jonge H, Lerut E, Verbeke K, Vanrenterghem Y. Tacrolimus dose requirements and CYP3A5 genotype and the development of calcineurin inhibitor-associated nephrotoxicity in renal allograft recipients. Ther Drug Monit. 2010 Aug;32(4):394-404. doi: 10.1097/FTD.0b013e3181e06818. PMID 20526235
- [Result] Naesens M, Lerut E, de Jonge H, Van Damme B, Vanrenterghem Y, Kuypers DR. Donor age and renal P-glycoprotein expression associate with chronic histological damage in renal allografts. J Am Soc Nephrol. 2009 Nov;20(11):2468-80. doi: 10.1681/ASN.2009020192. Epub 2009 Sep 17. PMID 19762492
- [Result] Evenepoel P, Lerut E, Naesens M, Bammens B, Claes K, Kuypers D, Vermeersch P, Meijers B, Van Damme B, Vanrenterghem Y. Localization, etiology and impact of calcium phosphate deposits in renal allografts. Am J Transplant. 2009 Nov;9(11):2470-8. doi: 10.1111/j.1600-6143.2009.02792.x. Epub 2009 Aug 14. PMID 19681815
- [Result] Naesens M, Li L, Ying L, Sansanwal P, Sigdel TK, Hsieh SC, Kambham N, Lerut E, Salvatierra O, Butte AJ, Sarwal MM. Expression of complement components differs between kidney allografts from living and deceased donors. J Am Soc Nephrol. 2009 Aug;20(8):1839-51. doi: 10.1681/ASN.2008111145. Epub 2009 May 14. PMID 19443638
- [Result] Evenepoel P, Van Den Bergh B, Naesens M, De Jonge H, Bammens B, Claes K, Kuypers D, Vanrenterghem Y. Calcium metabolism in the early posttransplantation period. Clin J Am Soc Nephrol. 2009 Mar;4(3):665-72. doi: 10.2215/CJN.03920808. Epub 2009 Mar 4. PMID 19261823
- [Result] Evenepoel P, Meijers BK, de Jonge H, Naesens M, Bammens B, Claes K, Kuypers D, Vanrenterghem Y. Recovery of hyperphosphatoninism and renal phosphorus wasting one year after successful renal transplantation. Clin J Am Soc Nephrol. 2008 Nov;3(6):1829-36. doi: 10.2215/CJN.01310308. Epub 2008 Oct 15. PMID 18922992
- [Result] Kuypers DR, de Jonge H, Naesens M, Vanrenterghem Y. Effects of CYP3A5 and MDR1 single nucleotide polymorphisms on drug interactions between tacrolimus and fluconazole in renal allograft recipients. Pharmacogenet Genomics. 2008 Oct;18(10):861-8. doi: 10.1097/FPC.0b013e328307c26e. PMID 18704002
- [Result] Naesens M, Lerut E, Damme BV, Vanrenterghem Y, Kuypers DR. Tacrolimus exposure and evolution of renal allograft histology in the first year after transplantation. Am J Transplant. 2007 Sep;7(9):2114-23. doi: 10.1111/j.1600-6143.2007.01892.x. Epub 2007 Jul 3. PMID 17608835
- [Result] Lerut E, Naesens M, Kuypers DR, Vanrenterghem Y, Van Damme B. Subclinical peritubular capillaritis at 3 months is associated with chronic rejection at 1 year. Transplantation. 2007 Jun 15;83(11):1416-22. doi: 10.1097/01.tp.0000266676.10550.70. PMID 17565313
- [Result] Evenepoel P, Naesens M, Claes K, Kuypers D, Vanrenterghem Y. Tertiary 'hyperphosphatoninism' accentuates hypophosphatemia and suppresses calcitriol levels in renal transplant recipients. Am J Transplant. 2007 May;7(5):1193-200. doi: 10.1111/j.1600-6143.2007.01753.x. Epub 2007 Mar 12. PMID 17359508
- [Result] Evenepoel P, Bammens B, Claes K, Kuypers D, Meijers BK, Vanrenterghem Y. Measuring total blood calcium displays a low sensitivity for the diagnosis of hypercalcemia in incident renal transplant recipients. Clin J Am Soc Nephrol. 2010 Nov;5(11):2085-92. doi: 10.2215/CJN.02460310. Epub 2010 Sep 9. PMID 20829423
- [Result] Kanaan N, Claes K, Devogelaer JP, Vanderschueren D, Depresseux G, Goffin E, Evenepoel P. Fibroblast growth factor-23 and parathyroid hormone are associated with post-transplant bone mineral density loss. Clin J Am Soc Nephrol. 2010 Oct;5(10):1887-92. doi: 10.2215/CJN.00950110. Epub 2010 Jul 15. PMID 20634326
- [Result] Claes K, Bammens B, Evenepoel P, Kuypers D, Coosemans W, Darius T, Monbaliu D, Pirenne J, Vanrenterghem Y. Troponin I is a predictor of acute cardiac events in the immediate postoperative renal transplant period. Transplantation. 2010 Feb 15;89(3):341-6. doi: 10.1097/TP.0b013e3181bc405e. PMID 20145526
- [Result] Naesens M, Heylen L, Lerut E, Claes K, De Wever L, Claus F, Oyen R, Kuypers D, Evenepoel P, Bammens B, Sprangers B, Meijers B, Pirenne J, Monbaliu D, de Jonge H, Metalidis C, De Vusser K, Vanrenterghem Y. Intrarenal resistive index after renal transplantation. N Engl J Med. 2013 Nov 7;369(19):1797-806. doi: 10.1056/NEJMoa1301064. PMID 24195547
- [Result] Khatri P, Roedder S, Kimura N, De Vusser K, Morgan AA, Gong Y, Fischbein MP, Robbins RC, Naesens M, Butte AJ, Sarwal MM. A common rejection module (CRM) for acute rejection across multiple organs identifies novel therapeutics for organ transplantation. J Exp Med. 2013 Oct 21;210(11):2205-21. doi: 10.1084/jem.20122709. Epub 2013 Oct 14. PMID 24127489
- [Result] De Vusser K, Lerut E, Kuypers D, Vanrenterghem Y, Jochmans I, Monbaliu D, Pirenne J, Naesens M. The predictive value of kidney allograft baseline biopsies for long-term graft survival. J Am Soc Nephrol. 2013 Nov;24(11):1913-23. doi: 10.1681/ASN.2012111081. Epub 2013 Aug 15. PMID 23949799
- [Result] Metalidis C, van Vuuren SH, Broekhuizen R, Lerut E, Naesens M, Bakker SJ, Wetzels JF, Goldschmeding R, Kuypers DR. Urinary connective tissue growth factor is associated with human renal allograft fibrogenesis. Transplantation. 2013 Sep 15;96(5):494-500. doi: 10.1097/TP.0b013e31829b07e1. PMID 23803600
- [Result] Naesens M, Kuypers DR, De Vusser K, Vanrenterghem Y, Evenepoel P, Claes K, Bammens B, Meijers B, Lerut E. Chronic histological damage in early indication biopsies is an independent risk factor for late renal allograft failure. Am J Transplant. 2013 Jan;13(1):86-99. doi: 10.1111/j.1600-6143.2012.04304.x. Epub 2012 Nov 8. PMID 23136888
- [Result] Lenain R, Dantan E, Giral M, Foucher Y, Asar O, Naesens M, Hazzan M, Fournier MC. External Validation of the DynPG for Kidney Transplant Recipients. Transplantation. 2021 Feb 1;105(2):396-403. doi: 10.1097/TP.0000000000003209. PMID 32108750
- [Result] Van Loon E, Senev A, Lerut E, Coemans M, Callemeyn J, Van Keer JM, Daniels L, Kuypers D, Sprangers B, Emonds MP, Naesens M. Assessing the Complex Causes of Kidney Allograft Loss. Transplantation. 2020 Dec;104(12):2557-2566. doi: 10.1097/TP.0000000000003192. PMID 32091487
- [Result] Senev A, Otten HG, Kamburova EG, Callemeyn J, Lerut E, Van Sandt V, Kuypers D, Emonds MP, Naesens M. Antibodies Against ARHGDIB and ARHGDIB Gene Expression Associate With Kidney Allograft Outcome. Transplantation. 2020 Jul;104(7):1462-1471. doi: 10.1097/TP.0000000000003005. PMID 31651716
- [Result] Heylen L, Thienpont B, Busschaert P, Sprangers B, Kuypers D, Moisse M, Lerut E, Lambrechts D, Naesens M. Age-related changes in DNA methylation affect renal histology and post-transplant fibrosis. Kidney Int. 2019 Nov;96(5):1195-1204. doi: 10.1016/j.kint.2019.06.018. Epub 2019 Jul 10. PMID 31530476
- [Result] Van Loon E, Gazut S, Yazdani S, Lerut E, de Loor H, Coemans M, Noel LH, Thorrez L, Van Lommel L, Schuit F, Sprangers B, Kuypers D, Essig M, Gwinner W, Anglicheau D, Marquet P, Naesens M. Development and validation of a peripheral blood mRNA assay for the assessment of antibody-mediated kidney allograft rejection: A multicentre, prospective study. EBioMedicine. 2019 Aug;46:463-472. doi: 10.1016/j.ebiom.2019.07.028. Epub 2019 Aug 1. PMID 31378695
- [Result] Zhang W, Yi Z, Keung KL, Shang H, Wei C, Cravedi P, Sun Z, Xi C, Woytovich C, Farouk S, Huang W, Banu K, Gallon L, Magee CN, Najafian N, Samaniego M, Djamali A, Alexander SI, Rosales IA, Smith RN, Xiang J, Lerut E, Kuypers D, Naesens M, O'Connell PJ, Colvin R, Menon MC, Murphy B. A Peripheral Blood Gene Expression Signature to Diagnose Subclinical Acute Rejection. J Am Soc Nephrol. 2019 Aug;30(8):1481-1494. doi: 10.1681/ASN.2018111098. Epub 2019 Jul 5. PMID 31278196
- [Result] Senev A, Lerut E, Van Sandt V, Coemans M, Callemeyn J, Sprangers B, Kuypers D, Emonds MP, Naesens M. Specificity, strength, and evolution of pretransplant donor-specific HLA antibodies determine outcome after kidney transplantation. Am J Transplant. 2019 Nov;19(11):3100-3113. doi: 10.1111/ajt.15414. Epub 2019 Jun 19. PMID 31062492
- [Result] Cippa PE, Liu J, Sun B, Kumar S, Naesens M, McMahon AP. A late B lymphocyte action in dysfunctional tissue repair following kidney injury and transplantation. Nat Commun. 2019 Mar 11;10(1):1157. doi: 10.1038/s41467-019-09092-2. PMID 30858375
- [Result] Coemans M, Van Loon E, Lerut E, Gillard P, Sprangers B, Senev A, Emonds MP, Van Keer J, Callemeyn J, Daniels L, Sichien J, Verbeke G, Kuypers D, Mathieu C, Naesens M. Occurrence of Diabetic Nephropathy After Renal Transplantation Despite Intensive Glycemic Control: An Observational Cohort Study. Diabetes Care. 2019 Apr;42(4):625-634. doi: 10.2337/dc18-1936. Epub 2019 Feb 14. PMID 30765434
- [Result] Senev A, Callemeyn J, Lerut E, Emonds MP, Naesens M. Histological picture of ABMR without HLA-DSA: Temporal dynamics of effector mechanisms are relevant in disease reclassification. Am J Transplant. 2019 Mar;19(3):954-955. doi: 10.1111/ajt.15234. Epub 2019 Jan 24. No abstract available. PMID 30582268
- [Result] Cippa PE, Sun B, Liu J, Chen L, Naesens M, McMahon AP. Transcriptional trajectories of human kidney injury progression. JCI Insight. 2018 Nov 15;3(22):e123151. doi: 10.1172/jci.insight.123151. PMID 30429361
- [Result] Yazdani S, Callemeyn J, Gazut S, Lerut E, de Loor H, Wevers M, Heylen L, Saison C, Koenig A, Thaunat O, Thorrez L, Kuypers D, Sprangers B, Noel LH, Van Lommel L, Schuit F, Essig M, Gwinner W, Anglicheau D, Marquet P, Naesens M. Natural killer cell infiltration is discriminative for antibody-mediated rejection and predicts outcome after kidney transplantation. Kidney Int. 2019 Jan;95(1):188-198. doi: 10.1016/j.kint.2018.08.027. Epub 2018 Nov 3. PMID 30396694
- [Result] Senev A, Coemans M, Lerut E, Van Sandt V, Daniels L, Kuypers D, Sprangers B, Emonds MP, Naesens M. Histological picture of antibody-mediated rejection without donor-specific anti-HLA antibodies: Clinical presentation and implications for outcome. Am J Transplant. 2019 Mar;19(3):763-780. doi: 10.1111/ajt.15074. Epub 2018 Sep 28. PMID 30107078
- [Result] Heylen L, Thienpont B, Naesens M, Busschaert P, Depreeuw J, Smeets D, Jochmans I, Monbaliu D, Pirenne J, Lerut E, Ghesquiere B, Kuypers D, Lambrechts D, Sprangers B. Ischemia-Induced DNA Hypermethylation during Kidney Transplant Predicts Chronic Allograft Injury. J Am Soc Nephrol. 2018 May;29(5):1566-1576. doi: 10.1681/ASN.2017091027. Epub 2018 Apr 2. PMID 29610404
- [Result] Azad TD, Donato M, Heylen L, Liu AB, Shen-Orr SS, Sweeney TE, Maltzman JS, Naesens M, Khatri P. Inflammatory macrophage-associated 3-gene signature predicts subclinical allograft injury and graft survival. JCI Insight. 2018 Jan 25;3(2):e95659. doi: 10.1172/jci.insight.95659. eCollection 2018 Jan 25. PMID 29367465
- [Result] De Vusser K, Pieters N, Janssen B, Lerut E, Kuypers D, Jochmans I, Monbaliu D, Pirenne J, Nawrot T, Naesens M. Telomere length, cardiovascular risk and arteriosclerosis in human kidneys: an observational cohort study. Aging (Albany NY). 2015 Oct;7(10):766-75. doi: 10.18632/aging.100814. PMID 26539975
- [Result] Naesens M, Lerut E, Emonds MP, Herelixka A, Evenepoel P, Claes K, Bammens B, Sprangers B, Meijers B, Jochmans I, Monbaliu D, Pirenne J, Kuypers DR. Proteinuria as a Noninvasive Marker for Renal Allograft Histology and Failure: An Observational Cohort Study. J Am Soc Nephrol. 2016 Jan;27(1):281-92. doi: 10.1681/ASN.2015010062. Epub 2015 Jul 7. PMID 26152270
- [Result] Delville M, Sigdel TK, Wei C, Li J, Hsieh SC, Fornoni A, Burke GW, Bruneval P, Naesens M, Jackson A, Alachkar N, Canaud G, Legendre C, Anglicheau D, Reiser J, Sarwal MM. A circulating antibody panel for pretransplant prediction of FSGS recurrence after kidney transplantation. Sci Transl Med. 2014 Oct 1;6(256):256ra136. doi: 10.1126/scitranslmed.3008538. PMID 25273097
- [Derived] Douwes RM, Gomes-Neto AW, Eisenga MF, Van Loon E, Schutten JC, Gans ROB, Naesens M, van den Berg E, Sprangers B, Berger SP, Navis G, Blokzijl H, Meijers B, Bakker SJL, Kuypers D. The association between use of proton-pump inhibitors and excess mortality after kidney transplantation: A cohort study. PLoS Med. 2020 Jun 15;17(6):e1003140. doi: 10.1371/journal.pmed.1003140. eCollection 2020 Jun. PMID 32542023